CLINICAL TRIAL: NCT05552807
Title: A Multicenter, Open Phase Ib Study to Evaluate the Efficacy and Safety of SCT-I10A in Combination With SCT200 or SCT200 in Combination With Paclitaxel/Docetaxel in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: SCT200 in Combination With SCT-I10A/Paclitaxel/Docetaxel in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT-I10A-B101; CTR20220916 (Registry Identifier: www.chinadrugtrials.org.cn); CTR20220917 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2022-06-22; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Squamous Carcinoma
Keywords: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 SCT200+SCT-I10A (Experimental): SCT200+SCT-I10A was given to patients who had failed previous platinum-based therapy. Among them, SCT200 was administered as 6 mg/kg/QW for 12 weeks and 8 mg/kg/Q2W maintenance by intravenous infusion; SCT-I10A was 200 mg/Q3W by intravenous infusion for no more than 2 years. Every 6 weeks is a treatment cycle. After the first dose, tumor assessment was performed every 6 weeks until the occurrence of PD, initiation of new antitumor therapy, withdrawal of informed consent, death, or loss of visit
  Interventions: Drug: SCT-I10A; Drug: SCT200
- Cohort 2-1 SCT200+SCT-I10A (Experimental): SCT200+SCT-I10A was given to patients who had failed previous platinum-based and immune checkpoint inhibitor therapy. Among them, SCT200 was administered as 6 mg/kg/QW for 12 weeks and 8 mg/kg/Q2W maintenance by intravenous infusion; SCT-I10A was 200 mg/Q3W by intravenous infusion for no more than 2 years. Every 6 weeks is a treatment cycle. After the first dose, tumor assessment was performed every 6 weeks until the occurrence of PD, initiation of new antitumor therapy, withdrawal of informed
  Interventions: Drug: SCT-I10A; Drug: SCT200
- Cohort 2-2 SCT200+paclitaxel/docetaxel (Experimental): SCT200+paclitaxel/docetaxel was given to patients who had failed previous platinum-based and immune checkpoint inhibitor therapy. Among them, SCT200 was administered as 6 mg/kg/QW for 12 weeks and 8 mg/kg/Q2W maintenance by intravenous infusion; paclitaxel was 80mg/m^2/QW by intravenous infusion; docetaxel was 75mg/m^2/Q3W. Every 6 weeks is a treatment cycle. After the first dose, tumor assessment was performed every 6 weeks until the occurrence of PD, initiation of new antitumor therapy, withdrawal of informed
  Interventions: Drug: SCT200; Drug: paclitaxel; Drug: docetaxel
- Cohort 3 SCT200+SCT-I10A (Experimental): SCT200+SCT-I10A was given to patients who have not received prior systemic chemotherapy. Among them, SCT200 was administered as 6 mg/kg/QW for 12 weeks and 8 mg/kg/Q2W maintenance by intravenous infusion; SCT-I10A was 200 mg/Q3W by intravenous infusion for no more than 2 years. Every 6 weeks is a treatment cycle. After the first dose, tumor assessment was performed every 6 weeks until the occurrence of PD, initiation of new antitumor therapy, withdrawal of informed
  Interventions: Drug: SCT-I10A; Drug: SCT200

INTERVENTIONS:
Drug: SCT-I10A — Administered intravenously
  Arms: Cohort 1 SCT200+SCT-I10A; Cohort 2-1 SCT200+SCT-I10A; Cohort 3 SCT200+SCT-I10A
Drug: SCT200 — Administered intravenously
Drug: paclitaxel — Administered intravenously
  Arms: Cohort 2-2 SCT200+paclitaxel/docetaxel
Drug: docetaxel — Administered intravenously
  Arms: Cohort 2-2 SCT200+paclitaxel/docetaxel

SUMMARY:
The study is to explore the efficacy and safety of SCT200 with SCT-I10A or SCT200 combined with paclitaxel/docetaxel in the treatment of recurrent/metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This multicenter, open phase Ib study focused on evaluating the objective response response rates of SCT200 in combination with SCT-I10A or SCT200 in combination with paclitaxel/docetaxel in patients with recurrent/metastatic head and neck squamous cell carcinoma who had previously received different treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed a written informed consent prior to screening;
2. Male or female, age ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Has histologically or cytologically confirmed head and neck squamous cell carcinoma;
5. Recurrent and/or metastatic HNSCC without indications for local radical treatment; Cohort 1: Patients who have received previous platinum-based therapy and experienced disease progression or toxic intolerance during or after treatment; Cohort 2: Patients who have received prior platinum-based therapy and immune checkpoint inhibitors and experienced disease progression or toxic intolerance during or after treatment; Cohort 3: Patients who have not received prior systemic chemotherapy but can receive chemotherapy as part of a multimodality treatment for patients with locally advanced HNSCC;
6. According to RECIST 1.1, there is at least one measurable lesion, for lesions previously treated with radiotherapy, may be selected as a target lesion only if the lesion has shown definite disease progression or persists more than 3 months after the end of radiotherapy;
7. The estimated survival period is ≥ 3 months;
8. Laboratory inspection: Blood test: neutrophils ≥1.5×10^9/L, hemoglobin ≥90g/L, platelets ≥75×10^9/L for cohort 1 and cohort 3, and platelets ≥100×10^9/L for cohort 2; liver function: Serum alanine transaminase (ALT) and serum aspartate aminotransferase (AST), ALT and AST ≤ 3 × ULN for those without liver metastases, ALT and AST ≤ 5 × ULN for those with liver metastases; total bilirubin (TBIL) ≤ 1.5 × ULN (Gilbert syndrome patients, ≤ 3 × ULN); Renal function: serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance (Ccr) ≥ 50 ml/min; Coagulation: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; Cardiac echocardiography: left ventricular ejection fraction (LVEF) ≥ 50%; Men and women of childbearing potential must agree that they must use contraception during the study period and for 6 months after the last study treatment; have a negative blood pregnancy test within 7 days prior to study enrollment and must non-breastfeeding

Exclusion Criteria:

1. Patients suitable for local radical treatment;
2. Histologically or cytologically confirmed nasopharyngeal or cutaneous squamous carcinoma;
3. Cohorts 1 and 3 previously treated with immune checkpoint inhibitors or treated with EGFR monoclonal antibodies (Immune-checkpoint inhibitors or EGFR monoclonal antibodies as multimodal therapy for locally advanced HNSCC were eligible if the last treatment was more than 6 months after disease progression);
4. Cohort 2 previously received EGFR monoclonal antibody (EGFR monoclonal antibodies as multimodal therapy for locally advanced HNSCC were eligible if the last treatment was more than 6 months after disease progression);
5. Cohort 2 previously received paclitaxel, albumin paclitaxel or paclitaxel liposomes, and received docetaxel, and both of these drugs failed to treat;
6. Previous immunotherapy with grade ≥3 irAE or grade ≥2 immune-associated myocarditis;
7. Other malignant neoplasm present within 5 years or concurrent with the current period, except cured cervical carcinoma in situ, non-melanoma skin cancer or other radically treated tumor/cancer with no signs of disease for at least 5 years;
8. Known peripheral neuropathy ≥ grade 2 according to the Common Terminology Criteria forAdverse Events(CTCAE v5.0) published by the National Cancer Institute (NCI);
9. Active central nervous system (CNS) metastases and/or carcinomatous meningitis;subjects with previously treated brain metastases may be enrolled in the study provided they are clinically stable for at least 2 weeks, have no evidence of new or expanding brain metastases, and have discontinued steroids at least 14 days prior to study drug administration. Stable brain metastases in this definition should be determined before the first dose of study drug. Subjects with asymptomatic brain metastases (i.e., no neurological symptoms, no need for corticosteroids, and no lesions >1.5 cm) may participate, but require periodic brain imaging at the the tumor lesion ;;
10. Subjects (except alopecia and hypothyroidism stabilized by hormone replacement therapy) who have not recovered from any toxicity and/or complications of previous surgery, chemotherapy or radiotherapy, i.e., who have not dropped to ≤ grade 1 (NCI CTCAE v5.0);
11. Any component of the study drug or formulation that has caused an allergic reaction, including a known grade ≥3 allergic reaction to other monoclonal antibody-based drugs;
12. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor therapy ≤ 4 weeks before the first dose, except palliative radiotherapy to the bone for pain relief; received nitrosourea or mitomycin C ≤ 6 weeks before the first dose; received fluorouracil and small molecule targeted drugs ≤ 2 weeks or ≤ 5 half-lives of the drug before the first dose; received Chinese medicine with anti-tumor indications ≤ 2 weeks before the first dose;
13. Received another unlisted clinical study drug or treatment ≤ 4 weeks prior to the first dose;
14. Major surgery ≤4 weeks prior to first dose or expected during this study;
15. Immunosuppressive drugs required ≤ 2 weeks prior to first dose or during the study period, excluding: a) intranasal, inhaled, topical glucocorticoids or topical glucocorticoid injections ; b) physiological doses of systemic glucocorticoids (≤ 10 mg/day prednisone or equivalent); c) short-term use of glucocorticoids for prophylaxis or treatment of non-autoimmune allergic diseases;
16. Subjects with known active, or with a history of autoimmune disease with a risk of relapse, or patients at high risk. However, the following patients are allowed to be enrolled: patients with type I diabetes who are stable with a fixed dose of insulin; autoimmune hypothyroidism who require only stable hormone replacement therapy; skin diseases that do not require systemic therapy;
17. Subjects with known history of interstitial lung disease, non-infectious pneumonia, or high suspicion of interstitial lung disease; subjects with previous drug-derived or radiological non-infectious pneumonia who are asymptomatic are allowed to be enrolled;
18. HIV positive, or other acquired or congenital immunodeficiency disease, or history of organ transplantation, or history of stem cell transplantation
19. HBsAg positive, and peripheral blood HBV DNA titer ≥ 2.5×10^3 copies/ml or ≥ 500 IU/ml; HCV antibody positive, and HCV-RNA above the lower limit of detection of the analytical method;
20. Active or uncontrollable infection requiring intravenous anti-infective therapy ≤ 2 weeks prior to the first dose;
21. Vaccination with live virus ≤ 4 weeks prior to first dose Seasonal influenza vaccine without live virus allowed;
22. Clinically uncontrollable third interstitial fluid that, in the judgment of the investigator, is not suitable for enrollment;
23. Known concomitant severe medical disease, such as NYHA III, IHD, or MI within 3 months prior to first dose, poorly controlled DM (fasting glucose ≥ 10 mmol/L) or poorly controlled hypertension despite drug therapy;
24. Medical or psychiatric history or history of laboratory abnormalities that may interfere with the interpretation of the results;
25. Subjects with alcohol or drug addiction;
26. Subjects deemed unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  ORR is defined as the proportion of subjects with complete response (CR) or partial response (PR) confirmed by the overall best response rate (assessed according to RECIST version 1.1).

SECONDARY OUTCOMES:
Disease control rate(DCR) | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  DCR is defined as the proportion of subjects who achieve best overall response of complete response (CR), partial response (PR) or stable disease (SD) according to RECIST version 1.1
Duration of response(DOR) | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  DOR is defined as the time from first response to first disease progression or death
Progression-free survival(PFS) | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  PFS is defined as the time between the date of first dose and the date of first documented disease progression (as assessed by RECIST version 1.1) or death from any cause.
Overall survival(OS) | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  OS is defined as the time from the date of first drug administration to death from any cause.
Correlation of PD-L1 expression level with efficacy and prognosis | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  For cohort1、2-1 and 3, evaluating correlation of PD-L1 expression level with efficacy and prognosis

OTHER OUTCOMES:
Occurrence of Study Treatment Related Adverse Events | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  Related adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0. An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product.
Immunogenicity | From date of the first dose until the date of first documented progression or date of receiving new antitumor therapy or date of withdraw informed consent or date of death from any cause, whichever came first，assessed up to 24 months
  Serum anti-SCT200 antibody and anti-SCT-I10A antibody levels before and after administration

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Ph.D, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin J, Qu S, Yang K, Zhang T, Bai Y, Wu J, Huang Y, Fang M, Liu X, Huang X, Chen N, Li Z, Li W, Zhang S, Zhang S, Hu G, Sun Y, Chen X, Liu Y, Jing S, Shen L, Chang Z, Xie L, Gai W, Zhou Q, Chen X, Yi J, Guo Y. Phase Ib study of SCT200 combined with paclitaxel or docetaxel in patients with recurrent or metastatic head and neck squamous cell carcinoma following platinum-based chemotherapy and PD-1 antibody. Cancer Lett. 2025 Mar 31;613:217513. doi: 10.1016/j.canlet.2025.217513. Epub 2025 Jan 30. PMID 39892704